CLINICAL TRIAL: NCT05074355
Title: Venetoclax and Azacitidine Combination Therapy for Patients With Accelerated or Blast Phase BCR-ABL Negative Myeloproliferative Neoplasm (VAAMP)
Brief Title: Study of Venetoclax and Azacitidine in Advanced BCR-ABL Negative Myeloproliferative Neoplasms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAAMP; 21-5928 (Other: University Health Network)
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacitidine and Venetoclax (Experimental): A treatment cycle is 28 days long.
  Azacitidine will be given by injection under the skin, once a day, for the first 6 days of every cycle.
  Venetoclax will be given orally, once a day, as follows at the discretion of their study doctors:
  Cycle 1:
  * Day 1 - 100 mg
  * Day 2 - 200 mg
  * Days 3 to 28 - 400 mg
  Cycle 2:
  * Participants with a response to the study drugs will continue taking 400 mg from Days 1 to 21, with no study drug from Days 22 to 28 during Cycle 2.
  * Participants who have not yet responded to the study drugs will continue taking 400 mg from Days 1 to 28 during Cycle 2.
  Cycle 3 and subsequent cycles:
  * Participants with a response to the study drugs will continue to take 400 mg from Days 1 to 21, with no study drug from Days 22 to 28.
  * Participants whose disease has not worsened will continue taking 400 mg from Days 1 to 28.
  * Participants have not responded to the study drugs will be withdrawn from the study.
  Interventions: Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Azacitidine is a hypomethylating agent that works by activating certain genes in the body to help cells mature and to kill abnormal bone marrow cells.
Drug: Venetoclax — Venetoclax is a drug that blocks a protein called B-cell lymphoma (BCL2) protein from working. BCL2 is a protein that helps control whether a cell lives or dies and is thought to help cancer cells to live. Blocking BCL2 is believed to help kill cancer cells.

SUMMARY:
The purpose of this research study is to look at how safe and useful a drug called azacitidine in combination with a drug called venetoclax, is in people with accelerated or blast phase BRC-ABL negative myeloproliferative neoplasms.

DETAILED DESCRIPTION:
All participants in this study will receive azacitidine and venetoclax.

This study will be done in multiple stages:

Safety Run-In Period - 7 participants will receive the study drugs to ensure that the combination is safe and tolerable.

Stage 1 - About 15 participants will receive the study drugs and will be evaluated to see whether they respond to the study drugs.

Stage 2 - If enough participants in Stage 1 respond to the study drugs, then Stage 2 will begin. During this stage, an additional 25 participants will take part in the study to further see if participants respond to the study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Ability to voluntarily provide written informed consent.
* Documented diagnosis per World Health Organization (WHO) 2016 criteria of BCR-ABL negative myeloproliferative neoplasms (MPN).
* Documented MPN transformation to accelerated phase (AP) or blast phase (BP) without prior blast reduction therapy for their AP/BP disease.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Adequate organ function.
* Must practice at least one reliable method of birth-control starting at least on cycle 1 day 1 until at least 90 days after the last dose of study drug.
* Female participants of childbearing potential must have a negative serum pregnancy test within 14 days prior to cycle 1 day 1.

Exclusion Criteria:

* History of allogeneic stem cell transplant for MPN.
* Previous treatment with venetoclax, navitoclax, azacytidine or other hypomethylating agents (HMA).
* White blood cell count >25 x 10^9/L.
* Current enrollment in another interventional study.
* Presence of any active uncontrolled infection such as bacterial or fungal infections progressing despite adequate antimicrobial treatment.
* Myocardial infarction in the preceding 3 months.
* Active human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV) infection.
* History of active malignancy in the previous 2 years.
* Any psychiatric illness or social circumstances or significant co-morbid conditions that may compromise study participation.
* Pregnant or breastfeeding women.
* Patients with known central nervous system (CNS) involvement with acute myeloid leukemia (AML) or CNS extramedullary hematopoiesis.
* Patients with t (15;17)
* Patients who have received strong and/or moderate CYP3A inducers within 7 days prior to the initiation of study treatment.
* Active COVID-19 infection.
* History of prior blast-reduction therapy for AP/BP-MPN.
* Preceding history MDS, chronic myelomonocytic leukemia (CMML), and other myelodysplastic syndromes (MDS)/MPN overlap syndromes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving complete remission (CR). | 3 years
Proportion of participants achieving complete remission with incomplete hematologic recovery (CRi). | 3 years
Proportion of participants achieving reversion to chronic myeloproliferative neoplasm (CMPN). | 3 years

SECONDARY OUTCOMES:
Average number of days from the first dose of azacytidine and venetoclax to the date of death. | 3 years
Average number of days from CR until relapse. | 3 years
Average number of days from CRi until relapse. | 3 years
Average number of days from CMPN until relapse. | 3 years
The proportion of patients proceeding to allogeneic stem cell transplantation in those eligible for transplantation. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Gupta, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada